CLINICAL TRIAL: NCT04544527
Title: The Risk Factors of Cardiovascular Disease in Elderly Diabetic Patients: A Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSE-202002
Record Dates: First submitted 2020-07-21; First posted 2020-09-10 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Complication Diabetic
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample, urinary sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the previous cohort studies focused on diabetes in China, there were few studies on elderly patients with diabetes. The aim of this prospective cohort study was to investigate the prevalence, management and nutritional status of elderly diabetic patients aged ≥65 years in Shanghai and Suzhou communities, and record the occurrence of endpoint events.

DETAILED DESCRIPTION:
This is a multicenter, observational, prospective cohort study.We plan to collect the baseline information in three years, and follow up every two years for at least 10 years. The study will enroll 5000 elderly diabetic patients aged ≥65 years and be conducted in Shanghai and Suzhou. The primary outcomes include MACE(major adverse cardiovascular events) , all-cause mortality, and chronic complications of diabetes and so on.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 65-100 years old;
* Patients who had been diagnosed with diabetes mellitus.

Exclusion Criteria:

* Patients with psychiatric disorders or impaired cognitive function;
* Patients who cannot or reject to sign the consent form.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This is a multicenter, observational, prospective cohort study.We plan to collect the baseline information in three years, and follow up every two years for at least 10 years. The study will enroll 5000 elderly diabetic patients aged ≥65 years and be conducted in Shanghai and Suzhou communities.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | Up to 10 years
  major adverse cardiovascular events,including the first occurrence of all-cause death, nonfatal myocardial infarction, or nonfatal stroke.
all-cause mortality | Up to 10 years
  All-cause mortality was confrmed through a combination of hospital medical records, telephone contacts with patients or family members, and death registration at the Xiangcheng Center for Disease Control and Prevention.

SECONDARY OUTCOMES:
chronic complications of diabetes | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (1):
- Xuejian Ni, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Anand SS, Dagenais GR, Mohan V, Diaz R, Probstfield J, Freeman R, Shaw J, Lanas F, Avezum A, Budaj A, Jung H, Desai D, Bosch J, Yusuf S, Gerstein HC; EpiDREAM Investigators. Glucose levels are associated with cardiovascular disease and death in an international cohort of normal glycaemic and dysglycaemic men and women: the EpiDREAM cohort study. Eur J Prev Cardiol. 2012 Aug;19(4):755-64. doi: 10.1177/1741826711409327. Epub 2011 May 6. PMID 21551215
- [Background] Hu Y, Ding M, Sampson L, Willett WC, Manson JE, Wang M, Rosner B, Hu FB, Sun Q. Intake of whole grain foods and risk of type 2 diabetes: results from three prospective cohort studies. BMJ. 2020 Jul 8;370:m2206. doi: 10.1136/bmj.m2206. PMID 32641435
- [Background] Li G, Zhang P, Wang J, Gregg EW, Yang W, Gong Q, Li H, Li H, Jiang Y, An Y, Shuai Y, Zhang B, Zhang J, Thompson TJ, Gerzoff RB, Roglic G, Hu Y, Bennett PH. The long-term effect of lifestyle interventions to prevent diabetes in the China Da Qing Diabetes Prevention Study: a 20-year follow-up study. Lancet. 2008 May 24;371(9626):1783-9. doi: 10.1016/S0140-6736(08)60766-7. PMID 18502303
- [Background] Huang ES, Liu JY, Moffet HH, John PM, Karter AJ. Glycemic control, complications, and death in older diabetic patients: the diabetes and aging study. Diabetes Care. 2011 Jun;34(6):1329-36. doi: 10.2337/dc10-2377. Epub 2011 Apr 19. PMID 21505211